CLINICAL TRIAL: NCT00192621
Title: A 3 Arm, Prospective Study to Compare the Effect of 6 Weeks Exposure to the Combination of Lopinavir (LPVr)/Combivir® (AZT/3TC) Versus Lopinavir Alone or Combivir® Alone in HIV-negative Healthy Subjects on the Development of Abnormalities of Lipid and Glucose Metabolism
Brief Title: Seronegatives and Metabolic Abnormalities Protocol 2 (SAMA002): Study to Compare the Effect of Kaletra and Combivir® in HIV-Negative Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: St Vincent's Hospital, Sydney (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Garvan Institute of Medical Research (Other); Prince of Wales Hospital, Sydney (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SAMA 002 Version 5; ACTR012605000661673
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections; Dyslipidemias; Glucose Metabolism Disorders; Metabolic Diseases; Lipodystrophy; Cardiovascular Disease
Keywords: HIV negative healthy subjects; Lipid metabolism; Glucose metabolism; Metabolic abnormality; Lipodystrophy; Cardiovascular disease; Treatment Naive; HIV
MeSH Terms: conditions — HIV Infections; Dyslipidemias; Glucose Metabolism Disorders; Metabolic Diseases; Lipodystrophy; Cardiovascular Diseases | interventions — lamivudine, zidovudine drug combination; Zidovudine; Lamivudine; lopinavir-ritonavir drug combination; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Combivir (zidovudine [AZT] / lamivudine [3TC])
Drug: Kaletra (lopinavir [LPVr])

SUMMARY:
This is a randomised study of the effect of treatment with Combivir (zidovudine [AZT] and lamivudine [3TC]) and Kaletra (lopinavir [LPVr]), alone and in combination, on the development of abnormalities in lipid and glucose metabolism in HIV negative healthy subjects.

DETAILED DESCRIPTION:
Antiretroviral medications, used to treat HIV infection, cause side effects. These include changes in the way that fat is laid down on the body. This results in fat loss from some parts of the body, with fat deposits at other sites, giving a characteristic look known as "HIV associated lipodystrophy" or HIVLD. With these changes, there are also abnormalities in glucose and fat metabolism (collectively termed metabolic abnormalities). In HIV negative populations, these metabolic changes are associated with an increased risk of developing cardiovascular disease (CVD). The aim of this study is to investigate if changes in the body's handling of fats and glucose occur with a short course of treatment in HIV negative subjects and if these correlate to an increased risk of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Be able to provide written consent to perform in the trial.
* HIV antibody negative and HIV DNA negative at time of entry to the study.

Exclusion Criteria:

* Any history of, or ongoing, mental or physical condition (including suspected or known diagnosis of ischaemic heart disease), which, in the opinion of the investigator, would impede the subject's ability to participate in the trial.
* History of type I or type II diabetes mellitus or previous treatment with antidiabetic medication.
* Prior use of testosterone, oestrogen, growth hormone or other oral glucocorticoid or anabolic steroid products within the previous six months.
* Alcohol or substance abuse which in the opinion of the investigator would affect the subject's ability to participate in the trial.
* Prior use of anti-retroviral agents (including protease inhibitors, nucleoside or non-nucleoside reverse transcriptase inhibitors, investigational antiretroviral agents or fusion inhibitors either in a previous study, as treatment or as part of post-exposure prophylaxis).
* Prior use of any retinoid-containing compound within the previous six months.
* Abnormal coagulation.
* Previous allergic reaction or known allergy to local anaesthetic.
* Previous use of psychotropic medications.
* Concomitant use of medications, including those metabolised by CYP3A4 enzyme system, which, in the opinion of the investigator, would affect the subject's ability to participate in all activities involved in the trial.
* Any grade-three laboratory abnormality recorded from screening bloods.
* Any grade-two laboratory abnormality recorded from screening bloods, which, in the opinion of the investigator, would impede the subject's ability to safely complete all study requirements.
* Gastrointestinal disorders, which may affect drug absorption.
* Any finding on screening clinical examination, which, in the opinion of the investigator, would impede the subject's ability to participate in the rest of the trial.
* Pregnancy
* Evidence of acute or chronic active hepatitis B virus infection by serology performed at baseline.
* Evidence of hepatitis C infection by serology performed at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine effect of 6 wks ART with LPVr and CBV, alone and in combination, in HIV negative healthy subjects with respect to changes from baseline in genes related to mitochondrial and lipid metabolism in adipocytes

SECONDARY OUTCOMES:
includes: To determine the effect of 6 wks of ART with LPVr and CBV in HIV negative subjects with respect to: changes from baseline in genes related to mitochondrial and lipid and glucose metabolism in monocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Carr, MD, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research.; David A Cooper, MD, Study Director — National Centre in HIV Epidemiology and Clinical Research.
Locations (1):
- St Vincents Hospital, Sydney, New South Wales, Australia

REFERENCES:
- See also: National Centre in HIV Epidemiology and Clinical Research Homepage — http://www.med.unsw.edu.au/nchecr/